CLINICAL TRIAL: NCT02747316
Title: Maternal Iron Absorption and Utilization and Iron Transfer to the Fetus During Pregnancy in Normal Weight and Overweight/Obese Women and the Effects on Infant Iron Status
Brief Title: Iron Absorption and Transfer to the Fetus During Pregnancy in Normal Weight and Overweight/Obese Women and the Effects on Infants Iron Status
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Isabelle Herter-Aeberli, Dr., Swiss Federal Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PIANO
Record Dates: First submitted 2016-01-08; First posted 2016-04-21 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Overweight; Obesity; Pregnancy
Keywords: Iron bioavailability; Hepcidin; Iron absorption
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotopically labeled test meal week of pregnancy 20 (Experimental)
  Interventions: Other: Stable iron isotope 57 (57Fe) labeled iron solution
- Isotopically labeled test meal week of pregnancy 30 (Experimental)
  Interventions: Other: Stable iron isotope 58 (58Fe) labeled iron solution

INTERVENTIONS:
Other: Stable iron isotope 57 (57Fe) labeled iron solution — test meal labeled with 12 mg 57Fe
  Arms: Isotopically labeled test meal week of pregnancy 20
Other: Stable iron isotope 58 (58Fe) labeled iron solution — test meal labeled with 12 mg 58Fe
  Arms: Isotopically labeled test meal week of pregnancy 30

SUMMARY:
Overweight and obesity causes low-grade systemic inflammation, which sharply increases risk for iron deficiency. Studies in our laboratory have shown that this is mainly the result of reduced dietary iron absorption because of increased hepcidin concentrations. During pregnancy, women have a large increase in iron needs because of the expansion of maternal blood volume and fetal needs. Iron deficiency anemia in infancy can impair cognitive development. Whether maternal adiposity impairs absorption and transfer of iron to the fetus, and thereby increases risk of iron deficiency in the mother and the infant is unclear.

DETAILED DESCRIPTION:
In obese subjects, hepcidin concentrations are increased and iron absorption is believed to be reduced, leading to iron deficiency over time. How all this will influence iron supply of the fetus in obese pregnancy has not been well investigated to date. Even if maternal and fetal iron uptakes are regulated separately, it is unclear to what extent maternal subclinical inflammation might influence this process. A small study by Dao et al. indicated that maternal-fetal iron transfer was impaired in obese pregnant women, possibly due to hepcidin up-regulation. In this study, both maternal BMI as well as hepcidin were negatively correlated with cord blood iron status. Maternal hepcidin and c-reactive protein were significantly higher and cord blood iron was significantly lower in the obese compared to the normal weight. Hepcidin was shown to have an effect on iron transfer across the placenta in the study by Young et al.: the transfer was increased in women with undetectable hepcidin at delivery compared to those with higher levels. As of now, clear associations between maternal BMI or maternal hepcidin concentration and fetal iron status were not shown.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with either normal pre-pregnancy BMI (BMI 18.5 - 24.9kg/kg2) or with overweight or obesity (BMI > 27.5kg/m2) before pregnancy (assessed based on data reported by the women at their first visit at the hospital)
* 18 to 45 years old
* singleton pregnancy
* week of pregnancy 14±3

Exclusion Criteria:

* underlying malabsorption disease
* chronic illness, which influences iron absorption
* inflammatory status other than obesity
* medical problems known to affect iron homeostasis
* smoking during pregnancy
* no regular use of medication, which influences iron absorption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | week 20 of pregnancy
  The fractional iron absorption from the first test meal will be calculated based on the shift of the iron isotopic ratios in the collected blood samples 14 days after administration of the isotopically labeled meal.
iron transfer from the mother to the fetus in cord blood/infant | delivery
  To determine the amount of iron transferred from the mother to the fetus
Fractional iron absorption | week 30 of pregnancy
  The fractional iron absorption from the second test meal will be calculated based on the shift of the iron isotopic ratios in the collected blood samples 14 days after administration of the isotopically labeled meal.
infants iron status | over the first six months of life
  infants iron status

SECONDARY OUTCOMES:
Change in plasma ferritin | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in plasma ferritin
Change in Hepcidin | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in Hepcidin
Change in transferrin receptor | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in transferrin receptor
Change in hemoglobin | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in hemoglobin
Change in c-reactive protein | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in c-reactive protein
Change in interleukin-6 | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in interleukin-6
Chage in alpha-1-acid glycoprotein | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Chage in alpha-1-acid glycoprotein
Change in retinol binding protein | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in retinol binding protein
Change in riboflavin | weeks of pregnancy 12, 18, 20, 28, 30, 36; 3 and 6 months after delivery
  Change in riboflavin
Assessment of children's iron needs within their first 2 years of life using an isotope dilution technique | Follow-up blood samples at 3, 6, 12, 18, 24 months after birth
  Assessment of children's iron needs within their first 2 years of life
Assessment of recovery of mother's iron Status after pregnancy using an isotope dilution technique | Follow-up blood samples at 3, 6, 12, 18, 24 months after delivery
  Assessment of recovery of mother's iron Status after pregnancy
infants iron status | over the first 24 months of life
  infants iron status

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Stoffel NU, Zimmermann MB, Cepeda-Lopez AC, Cervantes-Gracia K, Llanas-Cornejo D, Zeder C, Tuntipopipat S, Moungmaithong S, Densupsoontorn N, Quack Loetscher K, Gowachirapant S, Herter-Aeberli I. Maternal iron kinetics and maternal-fetal iron transfer in normal-weight and overweight pregnancy. Am J Clin Nutr. 2022 Apr 1;115(4):1166-1179. doi: 10.1093/ajcn/nqab406. PMID 34910118